CLINICAL TRIAL: NCT06382129
Title: A Phase III Randomized Controlled Clinical Study Comparing BL-B01D1 With Docetaxel in Patients With Unresectable Locally Advanced or Metastatic EGFR Wild-type Non-small Cell Lung Cancer After Failure of Anti-PD-1/PD-L1 Monoclonal Antibodies and Platinum-based Chemotherapy
Brief Title: A Study Comparing BL-B01D1 With Docetaxel in Patients With Unresectable Locally Advanced or Metastatic EGFR Wild-type Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-302
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BL-B01D1 (Experimental): Participants receive BL-B01D1 as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-B01D1
- Docetaxel (Experimental): Participants receive Docetaxel as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: BL-B01D1 — Administration by intravenous infusion for a cycle of 3 weeks.
  Other Names: iza-bren; izalontamab brengitecan; BMS-986507
  Arms: BL-B01D1
Drug: Docetaxel — Administration by intravenous infusion for a cycle of 3 weeks.
  Arms: Docetaxel

SUMMARY:
This trial is a registered phase III, randomized, open-label, multicenter study to evaluate the efficacy and safety of BL-B01D1 in patients with locally advanced or metastatic EGFR wild-type non-small cell lung cancer after failure of anti-PD-1/PD-L1 monoclonal antibodies and platinum-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent and follow the requirements of the protocol;
2. Age ≥18 years old;
3. Expected survival time ≥3 months;
4. Patients with histologically or cytologically confirmed locally advanced or metastatic EGFR wild-type non-small cell lung cancer;
5. Consent to provide archival tumor tissue samples or fresh tissue samples of primary or metastatic lesions within 3 years;
6. Must have at least one measurable lesion according to RECIST v1.1 definition;
7. ECOG 0 or 1;
8. Toxicity of previous antineoplastic therapy has returned to ≤ grade 1 defined by NCI-CTCAE v5.0;
9. No severe cardiac dysfunction, left ventricular ejection fraction ≥50%;
10. The organ function level must meet the requirements on the premise that blood transfusion is not allowed within 14 days before the screening period, and no cell growth factor drugs are allowed;
11. Urine protein ≤2+ or < 1000mg/24h;
12. For premenopausal women with childbearing potential, a pregnancy test must be performed within 7 days before the initiation of treatment, serum pregnancy must be negative, and must be non-lactating; All enrolled patients (male or female) were advised to use adequate barrier contraception throughout the treatment cycle and for 6 months after the end of treatment.

Exclusion Criteria:

1. Previous histological or cytological evidence of small cell or mixed small/non-small cell components;
2. Patients with EGFR L858R mutation, EGFR 19DEL mutation or EGFR T790M positive;
3. Chemotherapy, targeted therapy, biological therapy, etc., and palliative radiotherapy or antineoplastic therapy within 2 weeks before randomization;
4. Previous ADCs with TOPI inhibitors as toxins, antibodies/ADCs targeting EGFR and/or HER3;
5. History of severe heart disease or cerebrovascular disease;
6. Unstable thrombotic events requiring therapeutic intervention within 6 months before screening;
7. QT prolongation, complete left bundle branch block, III degree atrioventricular block, frequent and uncontrollable arrhythmia;
8. Active malignancy diagnosed within 3 years before randomization;
9. Hypertension poorly controlled by two antihypertensive drugs;
10. Patients with poor glycemic control;
11. A history of interstitial lung disease (ILD) requiring steroid therapy, or current ILD or grade ≥2 radiation pneumonitis, or suspicion of such disease on imaging during screening;
12. Complicated pulmonary diseases leading to clinically severe respiratory function impairment;
13. Patients with active central nervous system metastases;
14. Severe infection within 4 weeks before randomization; evidence of pulmonary infection or active pulmonary inflammation within 2 weeks before randomization;
15. Patients with massive or symptomatic effusions or poorly controlled effusions;
16. Imaging examination showed that the tumor had invaded or wrapped around the large blood vessels in the abdomen, chest, neck, and pharynx;
17. Severe unhealed wound, ulcer, or fracture within 4 weeks before signing the informed consent;
18. Subjects with clinically significant bleeding or obvious bleeding tendency within 4 weeks before signing the informed consent;
19. Patients with inflammatory bowel disease, extensive bowel resection history, immune enteritis history, intestinal obstruction or chronic diarrhea;
20. Have a history of allergy to recombinant humanized antibodies or any of the ingredients of BL-B01D1;
21. A history of autologous or allogeneic stem cell transplantation;
22. Human immunodeficiency virus antibody positive, active hepatitis B virus infection or hepatitis C virus infection;
23. A history of severe neurological or psychiatric illness;
24. Received other unmarketed investigational drug or treatment within 4 weeks before randomization;
25. Subjects who were scheduled to receive live vaccine or received live vaccine within 28 days before study randomization;
26. Any other circumstances in which the investigator considered it inappropriate to participate in the trial because of complications or other circumstances.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to approximately 24 months
  Overall survival (OS) is defined as the time between the subject's randomization date and subject's death.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 months
  Progression-free survival (PFS) as assessed by BIRC is defined as the time between the date subjects are randomized and the first observation of disease progression (based on BICR's image-based assessment) or death.
Objective Response Rate (ORR) | Up to approximately 24 months
  Objective response rate (ORR) is defined as the number of CR and PR in the treatment and control groups divided by the number of that group in the full analysis set (FAS).
Disease Control Rate (DCR) | Up to approximately 24 months
  Disease Control Rate (DCR) : Percentage of all randomized subjects who rated the best overall response (BOR) as complete response (CR), partial response (PR), and disease stabilization (SD) according to RECIST 1.1 criteria.
Duration of Response (DOR) | Up to approximately 24 months
  Duration of Response (DOR) : defined as the period from the date when tumor response is first recorded to the date when objective tumor progression is first recorded or the date of death.
Treatment Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-B01D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-B01D1.
Anti-drug antibody (ADA) | Up to approximately 24 months
  Frequency of anti-BL-B01D1 antibody (ADA) will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Wang, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China